CLINICAL TRIAL: NCT03422666
Title: Investigating the Plasma Lipoprotein Response to a Single Subcutaneous Dose of Analogue Glucagon-like Peptide-2 in Humans
Brief Title: Plasma Lipoprotein Response to Glucagon-like Peptide-2
Acronym: GLP-2 Plasma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-6368.1
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2021-04

CONDITIONS: Hyperlipidemias
Keywords: Intestinal lipoprotein; Gut Peptide; Chylomicrons
MeSH Terms: conditions — Hyperlipidemias | interventions — teduglutide

STUDY DESIGN:
Intervention Model Description: On visits 3 & 4, participants will receive either teduglutide or placebo, in random order, 5 hours after a high-fat drink
Who Masked: Participant
Masking Description: Single-blinded study with participant blinded to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teduglutide (Experimental): Teduglutide, up to 0.05mg/kg, subcutaneous, single dose
  Interventions: Drug: Teduglutide
- Placebo (Placebo Comparator): Placebo, subcutaneous, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teduglutide — Teduglutide
  Arms: Teduglutide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Some of the fat (triglyceride) from the food humans eat gets stored in the bowel. This triglyceride can then be released into the blood when another meal is consumed or in response to hormones. How the gut hormone glucagon-like peptide-2 (GLP-2) releases the triglyceride from the gut is not known. The research team in this study is interested in finding out how teduglutide (a degradation resistant form of GLP-2) releases stored triglyceride from the gut by evaluating how blood lipoproteins respond to teduglutide in healthy individuals.

DETAILED DESCRIPTION:
The lipoprotein response will be performed in 15 healthy individuals recruited by newspaper advertisements. Each subject will be their own control, receiving both placebo and teduglutide, administered on separate occasions. A member of the study team will explain the study in detail on visit 1, and if the individual is interested in participating, informed consent will be obtained and preliminary screening will occur on visit 2. On visit 3 & 4 participants will receive a high fat liquid meal after an overnight fast. Hourly blood samples will be taken for 5 hours, followed by randomized assignment to receive either subcutaneous placebo or teduglutide at visit 3 and the opposite treatment at visit 4. Following the injection, blood samples will be taken every 15 minutes for the first hour and every 30 minutes for the subsequent 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 60 years.
* Body mass index 20 to 27 kg/m2

Exclusion Criteria:

* Patients with active inflammatory bowel disease
* Patients with pre-existing Celiac disease, exocrine pancreatic insufficiency or small bowel malabsorption
* Patients with active bowel malignancy
* Patients with diabetes mellitus or known/ suspected motility disorders of the gut
* Patients with decompensated liver disease
* Patients on ezetimibe or bile acid sequestrants
* Patients who are pregnant or breastfeeding.
* Patients with renal disease.
* Patients on benzodiazepine.
* Unstable cardiac or respiratory disease
* Any changes to medication in the preceding month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Lipoprotein response to teduglutide | 8 hours
  To quantify the plasma lipoprotein response to teduglutide (GLP-2 analogue) injection in healthy individuals

CONTACTS AND LOCATIONS:
Overall Officials: Gary Lewis, MD, Principal Investigator — UHN
Locations (1):
- Toronto General Hopital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No